CLINICAL TRIAL: NCT00972413
Title: Cone Beam Computed Tomography for Breast Imaging and IV Contrast Enhanced Cone Beam Computed Tomography Breast Imaging
Brief Title: Cone Beam Computed Tomography for Breast Imaging
Acronym: CBCTBI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Koning Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KBCT-001
Record Dates: First submitted 2009-09-03; First posted 2009-09-07 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Breast Cancer
Keywords: breast cancer; cone beam computed tomography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group I (Experimental)
  Interventions: Radiation: Computed Tomography
- Group II (Experimental)
  Interventions: Radiation: Computed Tomography
- Group III (Experimental)
  Interventions: Radiation: Computed Tomography

INTERVENTIONS:
Radiation: Computed Tomography — In Group I, twelve CBCT studies will be performed. The objectives will be to illustrate the capacity of CBCT to image the breast in its entirety as compared with the gold standard mammographic exam.
  Arms: Group I
Radiation: Computed Tomography — In Group II , at least fifty (50) study participants, who are categorized as BI-RADS® 4, 5 based on prior diagnostic work-up and are also scheduled for breast biopsy of a lesion, will undergo a breast CBCT specifically designed to image the breast.
  Arms: Group II
Radiation: Computed Tomography — In Group III, at least 30 study subjects, who are categorized as BI-RADS® 4, 5 based on prior diagnostic work-up and are also scheduled for breast biopsy of a lesion, will undergo a unilateral intravenous (IV) CE CBCT of the involved breast.
  Arms: Group III

SUMMARY:
The primary aim of this study is to investigate the use of cone beam computed tomography (CBCT) for breast imaging in the diagnostic setting by providing a compelling body of evidence incorporating both non-contrast and contrast enhanced CBCT in the study protocol. The goal is to accumulate a body of evidence to provide data to incorporate CBCT into the diagnostic work-up of breast lesions.

ELIGIBILITY:
Inclusion Criteria:

Group I:

* Are at least 40 years of age of any ethnicity
* Had a mammogram, read as BI-RADS® 1 or 2
* Will undergo study imaging no later than four weeks from date of mammogram.
* Is able to undergo informed consent.

Group II:

* Are at least 40 years of age of any ethnicity
* Had a routine mammogram, read as BI-RADS® 4 or 5
* Are scheduled for breast biopsy
* Will undergo study imaging no later than four weeks from date of mammogram, prior to breast biopsy.
* Is able to undergo informed consent.

Group III:

* Are at least 40 years of age of any ethnicity
* Had a routine mammogram, read as BI-RADS® 4 or 5
* Are scheduled for breast biopsy
* Will undergo study imaging no later than four weeks from date of mammogram, prior to breast biopsy.
* Is able to undergo informed consent.

Exclusion Criteria:

Group I and Group II:

* Pregnancy
* Lactation
* Subjects with physical limitations that may prohibit resting prone on the exam table, such as, but not limited to: frozen shoulder, recent heart surgery, pace maker.
* Subjects who are unable to tolerate study constraints.
* Subjects who have received radiation treatments to the thorax for malignant and nonmalignant conditions, such as (but not limited to)

  * Treatment for enlarged thymus gland as an infant
  * Irradiation for benign breast conditions, including breast inflammation after giving birth
  * Treatment for Hodgkins disease
* Subjects who have participated in a prior breast clinical trial that gave additional radiation dose, such as an additional mammogram.
* Subjects who have received large numbers of diagnostic x-ray examinations for monitoring of disease such as (but not limited to)

  * Tuberculosis
  * Severe scoliosis

Group III:

* Pregnancy
* Lactation
* Subjects with physical limitations that may prohibit resting prone on the exam table, such as, but not limited to: frozen shoulder, recent heart surgery, pace maker.
* Subjects who are unable to tolerate study constraints.
* Subjects who have received radiation treatments to the thorax for malignant and nonmalignant conditions, such as (but not limited to)

  * Treatment for enlarged thymus gland as an infant
  * Irradiation for benign breast conditions, including breast inflammation after giving birth
  * Treatment for Hodgkins disease
* Subjects who have participated in a prior breast clinical trial that gave additional radiation dose, such as an additional mammogram.
* Subjects who have received large numbers of diagnostic x-ray examinations for monitoring of disease such as (but not limited to)

  * Tuberculosis
  * Severe scoliosis
* Allergy or previous reaction to iodinated contrast material
* History of renal dysfunction/kidney disease
* Long standing diabetes mellitus
* Multiple myeloma
* Dehydration
* History of nephrotoxic medication use
* Hyperthyroidism
* Diabetic patients on Metformin
* Pheochromocytoma
* Sickle Cell Disease

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2008-06; Primary Completion 2010-01 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
The study's intent is to provide compelling data to illustrate the potential contribution of CBCT for breast imaging, not to generate statistically significant data. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Posy Seifert, D.O., Principal Investigator — Elizabeth Wende Breast Care, LLC
Locations (1):
- Elizabeth Wende Breast Care, Rochester, New York, United States